CLINICAL TRIAL: NCT05594654
Title: A Digital Respiratory Ecosystem for People Living With Asthma: Mixed Methods
Brief Title: A Digital Respiratory Ecosystem for People Living With Asthma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asthma Research Group Windsor-Essex Inc (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Christopher Licskai, Principle Investigator, Asthma Research Group Windsor-Essex Inc
Other Study IDs: ARGI-001
Record Dates: First submitted 2022-05-10; First posted 2022-10-26 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Smart Phone Application — Breathe is an app that can be used by people with asthma to promote collaborative self-management. It is a platform that empowers patients to self-manage their condition. Breathe helps patients detect when they might be exacerbating or adequately controlled based on symptoms entered by the user into the application. The application then feeds these symptoms through a rules-based algorithm that identifies the early onset of an exacerbation, based on the user's "zone of control" or action plan. It also stores the patient's self-management action plan and gives them relevant instructions when it sees that their symptoms are getting better or worse. These instructions are delivered through a chatbot that provides information, support, and education to the patient through a friendly, human-like text message conversation.
  Other Names: Breathe Application

SUMMARY:
The purpose of this pilot study is to establish the feasibility and acceptability of a digital respiratory ecosystem ("Breathe"), that incorporates an acoustic adherence algorithm, asthma/COPD differentiation classification algorithm, a smart inhaler cap, a digital spirometer, and a real-time air quality database to support people living with asthma to better manage their disease and derive personal and clinical value. Through this study, 30 adults will be asked to use Breathe as a way to monitor and manage their asthma symptoms over a 12-week period.

DETAILED DESCRIPTION:
Asthma is one of the most common respiratory diseases globally and its prevalence is increasing. On average, 7.8% of Canadians were diagnosed with asthma in 2019. The direct and indirect impacts of asthma affects individuals physically, emotionally, and socially. As a chronic disease, the health and economic cost of asthma continues to grow. Asthma is a leading cause of disability and premature mortality in Canada. By 2030, it is estimated that asthma will cost Canadians more than $4 billion annually. Due to severe asthma exacerbations, there have been over 60,000 emergency room visits in 2019. However, these occurrences could have been averted with effective prevention and management measures. Several studies have indicated that only 50% of asthma patients in Canada are able to control the disease effectively.

In 2014, a digital respiratory application called Breathe was developed to support Canadians living with asthma. The first iteration of Breathe was developed as a self-monitoring and self-management web- and mobile-based application. Patients had access to their personal health information and electronic health records in order to understand their asthma care plan. The application shared asthma-related data with caregivers and health care providers to enhance the patient's asthma care. The features of the application were an action plan, daily and weekly symptom assessments, medication details, trend analyses, and alerting the patient of modifications in their asthma control zone.

Breathe 2.0 was adapted into a multi-functional iOS platform that offers dynamic and passive input through a chatbot, insights, predictions, and preventative measures to the user. These features included self-management asthma action plan, daily and weekly symptom assessment, and medication information, rich visualization of user data for review and trend analysis, and alerting functions to warn users of changes in their asthma control zone. In 2018, a randomized controlled trial of 138 patients was conducted with Breathe 2.0 to evaluate patient outcomes. This study concluded that individuals with asthma reported good usability and high satisfaction levels through the System Usability Scale. Furthermore, patients had high confidence in the platform's assessment of asthma control and the respective recommendations.

While Breathe 2.0 gave patients a platform to view and share information related to their symptoms, the app was cumbersome and required participants to manually enter their information; did not capture medication adherence which is an essential part of asthma symptom management, and did not incorporate spirometry insights into the algorithmic determination of asthma control.

This updated version of Breathe will be able to:

* Aid physicians in confirming the patient's diagnosis of Asthma or COPD through the use of the Asthma COPD differentiation classification algorithm
* Encourage and track medication adherence for both maintenance medications and use of rescue medications
* Educate users to recognize and manage their symptoms, and ensure they are adequately controlled
* Provide and promote the use of a customized action plan
* Monitor the use and effectiveness of the action plan
* Provide robust and granular weather, air quality and pollen forecasts to assist patients in identifying potential environmental triggers
* Introduce daily Spirometry testing and the importance of tracking and understanding Spirometry values and a "best number"

In this pilot study, investigators aim to evaluate the feasibility and acceptability of Breathe as a self-monitoring and self-management tool for asthma. Through this study, investigators seek to identify barriers to adoption and areas for improvement of the Breathe technology and to create a service model that will guide the implementation of this technology, allowing for a more widespread use of the intervention to be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Between 18 - 80 years of age
* Have a clinical diagnosis of asthma
* Received Global Initiative of Asthma (GINA) Step 3-5 asthma therapies to manage moderate to severe asthma
* Have been using Enerzair or Atectura maintenance medications for at least 2 weeks
* Currently prescribed a salbutamol rescue medication administered through a pressurized metered dose inhaler (MDI)
* Adequate English ability to complete study activities as determined by the study staff
* Own an iPhone that is compatible with the intervention (i.e. iPhone 7 or above, iOS 14 or above, and connected to an active data plan)

Exclusion Criteria:

* They are already under the care of a certified respiratory educator for uncontrolled asthma management
* They have another pulmonary disease (e.g. COPD) that will impact their ability to use the intervention as intended (as deemed by the recruiting clinician)
* They have a medical condition that would limit their ability to self-manage their asthma (as deemed by the recruiting clinician)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty adults with a clinical diagnosis of asthma will be enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Engagement | Measured at 12-weeks
  Number of unique days patient used the Breathe app
Component Engagement | Measured at 12-weeks
  Assess by how often patients are using the different components of the breathe app.
Technical Issues | Measured at 12-weeks
  Assess the number of technical issues reported.

SECONDARY OUTCOMES:
Changes in Patient's Inhaler Technique | Measured at continuously over 12- weeks; at baseline and at 12-weeks
  Assessed by the number of inhaler technique errors detected by in-app tool, in-app audio recording of medication inhaler and formal assessment of inhaler technique done in clinic.
Changes in the quality of home spirometry | Measured continuously for 12-weeks and at 12-weeks
  Assessed by the number of failed spirometry tests detected by in-app digital spirometer, formal assessment of unsupported test completed at clinic and patient experience feedback survey.
Medication Adherence | Measured at 12-weeks
  Assessed by the electronic measures of adherence through the Breathe application.
Changes to asthma-related quality of life | Measured at Baseline and 12- weeks
  Assessed by the Mini Asthma Quality of Life questionnaire. This questionnaire contains 15-questions that asses the quality of health-related well-being for patients living with asthma. The minimal value is 15 and the maximum value is 105. The higher score represents a better quality of life
Changes to Asthma Control | Measured at Baseline, 12-weeks and continuously for 12-weeks
  Assessed by the Asthma Control Questionnaire. The Asthma Control Questionnaire is a 6-item instrument used to quantify a patient's asthma control. The minimal value is 0 and the maximum value is 36. A higher score represents poorer asthma control.
Diagnostic Alignment | Measured at 12-weeks
  Assessed by comparing the breathe application diagnostic output, the patient's historical clinical diagnosis of asthma and the most recent clinical diagnosis.
Changes to Satisfaction with Care | Measured at baseline and at 12-weeks
  Assessed by the Satisfaction of Care questionnaire. This questionnaire contains 3 questions used to quantify experience and acceptability of the Breathe ecosystem. The minimal value is 3 and the maximum value is 15. A higher score represents high user satisfaction.
Changes to Treatment Behaviour | Measured at Baseline and 12-weeks
  Assessed by the Observed Treatment Behaviour Questionnaire. This questionnaire is a 43-item instrument that quantifies a patient's attitude towards their asthma and treatment. The minimum value is 43 and the maximum value is 215. A higher score represents poorer attitude toward asthma and treatment.
Changes to patient's healthcare utilization | Measured at Baseline and 12- weeks
  Assessed by the number of urgent asthma-related health care visits following an asthma exacerbation.
Maintenance Medication Adherence | Measured at 12-weeks
  Assessed by formal dose counting of maintenance medication done in clinic at study end.
Rescue Medication Use | Measured at 12-weeks
  Assessed by the number of rescue inhaler uses detected by a peripheral inhaler component.
Asthma Control | Measured at 12-weeks
  Percentage of time spent across asthma action plan zones of control.

CONTACTS AND LOCATIONS:
Locations (1):
- Asthma Research Group Windsor Essex County Inc, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Findings from the study will be published and shared through open accessed peer review journals and scientific conferences within the digital health and cancer respective fields. Results will be shared in aggregate.